CLINICAL TRIAL: NCT00976950
Title: A Post Marketing Surveillance Study Assessing the Long-term Efficacy and Safety of Tipranavir (Aptivus®) Co-administered With Low-dose Ritonavir in Treatment Experienced Patients With HIV-1 Infection in the Daily Clinical Practice.
Brief Title: A Post Marketing Surveillance Study Assessing the Long-term Efficacy and Safety of Aptivus Co-administered With Low-dose Ritonavir in Treatment Experienced Patients With HIV-1 Infection in the Daily Clinical Practice.
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1182.147
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2012-08-16 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with HIV-1 infection
  Interventions: Drug: Tipranavir; Drug: ritonavir

INTERVENTIONS:
Drug: Tipranavir
Drug: ritonavir — low-dose

SUMMARY:
The aim of this trial is to evaluate the safety and virological and immunological efficacy of Aptivus in treatment-experienced patients with advanced HIV-1 infection who had developed resistance to more than one protease inhibitor.

ELIGIBILITY:
Inclusion criteria:

1. HIV-1 infected patients who are treatment experienced and infected with HIV-1 strains resistant to more than one protease inhibitor and no other therapeutic options.
2. The inclusion criteria follow the same criteria which are describe in the newest SPC

Exclusion criteria:

The exclusion criteria follow the same criteria which are describe in the newest SPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (20):
- Romania (20):
  - Boehringer Ingelheim Investigational site 9, Arad
  - Boehringer Ingelheim Investigational site 13, Bacau
  - Boehringer Ingelheim Investigational site 17, Brasov
  - Boehringer Ingelheim Investigational site 18, Brasov
  - Boehringer Ingelheim Investigational site 19, Brasov
  - Boehringer Ingelheim Investigational site 1, Bucharest
  - Boehringer Ingelheim Investigational site 2, Bucharest
  - Boehringer Ingelheim Investigational site 3, Bucharest
  - Boehringer Ingelheim Investigational site 4, Bucharest
  - Boehringer Ingelheim Investigational site 5, Bucharest
  - Boehringer Ingelheim Investigational site 6, Bucharest
  - Boehringer Ingelheim Investigational site 7, Bucharest
  - Boehringer Ingelheim Investigational site 8, Bucharest
  - Boehringer Ingelheim Investigational site 16, Constanța
  - Boehringer Ingelheim Investigational site 11, Craiova
  - Boehringer Ingelheim Investigational site 12, Craiova
  - Boehringer Ingelheim Investigational site 15, Galati
  - Boehringer Ingelheim Investigational site 20, Tg.Mures
  - Boehringer Ingelheim Investigational site 10, Timișoara
  - Boehringer Ingelheim Investigational site 14, Vaslui

RESULTS

PARTICIPANT FLOW:
Groups:
- Aptivus and Ritonavir: TPV/r means Treated with Tipranavir (Aptivus) 500mg twice daily and low-dose ritonavir
Period: Overall Study
Arm/Group | Aptivus and Ritonavir
Started | 42
Completed | 36
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Events with no relationship to Aptivus | 3

BASELINE CHARACTERISTICS:
Arm/Group | Aptivus and Ritonavir
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — Age is available for 41 patients.
  years | 25.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 23
Baseline HIV RNA values [Number; unit: Participants]
  <= 50 copies/ml | 0
  51 - <1,000 copies/ml | 1
  1,000 - <10,000 copies/ml | 5
  10,000 - <100,000 copies/ml | 13
  100,000 - <1,000,000 copies/ml | 12
  >= 1,000,000 copies/ml | 0
  Missing | 11
Baseline CD4+ count [Number; unit: Participants]
  <= 50 cells/mm^3 | 2
  51 - <251 cells/mm^3 | 19
  251 - <451 cells/mm^3 | 13
  >= 451 cells/mm^3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Adverse Events (AE)
Description: Any type of adverse events
Time Frame: 48 weeks
Population: Treated set (TS), defined as patients treated with Aptivus
Measure: Number; unit: Participants
Arm/Group | Aptivus and Ritonavir
Number analyzed (Participants) | 42
Participants
  Patients with any adverse events | 6
  Patients with any serious adverse events | 1
  Patients with AE leading to discontinuation | 4
  Patients with hepatic adverse events | 1
  Patients with dyslipidemia | 2

2. Secondary Outcome: Virologic Response
Description: Virologic response is defined as HIV viral load of < 50 copies/mL before week 48 and without subsequent rebound or change of ARV therapy prior to week 48. A rebound is defined by two consecutive measurements of VL >= 50 copies/ml, at least two weeks apart, after two consecutive measurements of VL< 50 copies/ml. Because of many missing data concerning the viral load, the virologic response could be determined only for four patients.
Time Frame: 48 weeks
Population: Treated set (TS), defined as patients treated with Aptivus
Measure: Number; unit: Number of participants
Arm/Group | Aptivus and Ritonavir
Number analyzed (Participants) | 42
Number of participants
  Virologic response - Yes | 0
  Virologic response - No | 4
  Virologic response - Missing | 38

3. Secondary Outcome: Change in CD4+ Cell Count From Baseline at Week 48
Time Frame: 48 weeks
Population: Treated set with with non-missing data at the visit
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Aptivus and Ritonavir
Number analyzed (Participants) | 28
cells/mm^3 | 85.8 (29.6)

ADVERSE EVENTS:
Groups:
- Aptivus and Ritonavir: ARV means Treated with Tipranavir (Aptivus) 500mg twice daily and low-dose ritonavir
Arm/Group | Aptivus and Ritonavir
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 0/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aptivus and Ritonavir (N=42)
Pulmonary tuberculosis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.